CLINICAL TRIAL: NCT02715635
Title: A Double-blind, Randomised, Placebo-controlled Parallel Study to Investigate the Effect of Dietary Nitrate on a Model of Vascular Dysfunction in Healthy Volunteers
Brief Title: Influence of Dietary Nitrate on Vascular Dysfunction and Inflammation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Amrita Ahluwalia, Director of The William Harvey Research Institute, Prof of Vascular Pharmacology, Queen Mary University of London
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 15/LO/0789
Record Dates: First submitted 2016-03-16; First posted 2016-03-22 (Estimated); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Typhoid-Paratyphoid Vaccines; Vi polysaccharide vaccine, typhoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitrate-rich beetroot juice (Active Comparator): Biological: Typhoid vaccine The typhoid vaccine is composed of purified polysaccharide from S. typhi capsule 25 micrograms contained in 0.5 ml solution Other Name: Typhim Vi®
  Dietary Supplement: Concentrate beetroot Juice 140 ml containing ~8 mmol of inorganic nitrate
  Interventions: Biological: Typhoid vaccine; Dietary Supplement: Concentrate beetroot Juice
- Nitrate-deplete beetroot juice (Placebo Comparator): Biological: Typhoid vaccine The typhoid vaccine is composed of purified polysaccharide from S. typhi capsule 25 micrograms contained in 0.5 ml solution Other Name: Typhim Vi®
  Dietary Supplement: Concentrate beetroot Juice 140 ml which is nitrate-depleted
  Interventions: Biological: Typhoid vaccine; Dietary Supplement: Concentrate beetroot Juice (Placebo)

INTERVENTIONS:
Biological: Typhoid vaccine — The typhoid vaccine is composed of purified polysaccharide from S. typhi capsule 25 micrograms contained in 0.5 ml solution
  Other Names: Typhim Vi®
Dietary Supplement: Concentrate beetroot Juice — 140 ml containing ~8 mmol of inorganic nitrate
  Arms: Nitrate-rich beetroot juice
Dietary Supplement: Concentrate beetroot Juice (Placebo) — 140 ml which is nitrate-depleted
  Arms: Nitrate-deplete beetroot juice

SUMMARY:
The principal research objective is to determine whether inorganic nitrate in the form of beetroot juice compared to placebo control prevents the systemic inflammation that underlies typhoid vaccine-induced endothelial dysfunction

DETAILED DESCRIPTION:
We wish to determine in a prospective manner whether inorganic nitrate affects the endothelial dysfunction induced by systemic inflammation. At baseline we will measure flow-mediated dilatation (FMD) and peripheral augmentation index, as well as aortic stiffness, as measured by pulse wave velocity (PWV). Volunteers will then receive ~8 mmols of dietary nitrate or nitrate free placebo juice once daily for 6 days. After this, depending on availability, volunteers will receive a typhoid vaccine Typherix®, GlaxoSmithKline UK or Typhim Vi ™, AAH Pharmaceuticals Ltd). This vaccine generates a mild systemic inflammation that is associated with vascular dysfunction. All vascular function measures will be repeated at 8 hours and 32 hours after vaccine administration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers
2. Aged 18-45
3. Volunteers who are willing to sign the consent form.
4. Normal resting blood pressure (<140/90 mmHg)

Exclusion Criteria:

1. Healthy subjects unwilling to consent
2. Pregnant, or any possibility that a subject may be pregnant unless in the latter case a pregnancy test is performed with a negative result
3. History of any serious illnesses, including recent infections or trauma
4. Subjects taking systemic medication (other than the oral contraceptive pill)
5. Subjects with self-reported use of mouthwash or tongue scrapes
6. Subjects with recent (3 months) or current antibiotic use
7. Subjects with a history, or recent treatment of (within last 3 months) any oral condition (excluding caries), including gingivitis, periodontitis and halitosis
8. Subjects with a history of typhoid vaccination in the last 6 months
9. Subjects with any history of a blood-borne infectious disease such Hepatitis B or C virus, or HIV

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Flow mediated dilatation | Day 1, Day 7 (8 hours post typhoid vaccine), Day 8 (32 hours post typhoid vaccine)
  Comparison of change in FMD from baseline after typhoid vaccination following inorganic nitrate versus placebo supplementation
Plasma nitrite concentration | Day 1, Day 7 (8 hours post typhoid vaccine), Day 8 (32 hours post typhoid vaccine)
  Comparison of change in plasma nitrite concentration following inorganic nitrate versus placebo supplementation

SECONDARY OUTCOMES:
Markers of acute inflammation | Day 1, Day 7 (8 hours post typhoid vaccine), Day 8 (32 hours post typhoid vaccine)
  Comparison of change in peripheral markers of inflammation and leucocyte count following nitrate versus placebo supplementation
Pulse wave velocity | Day 1, Day 7 (8 hours post typhoid vaccine), Day 8 (32 hours post typhoid vaccine)
  Comparison of change in PWV from baseline after typhoid vaccination following nitrate versus placebo supplementation
Platelet reactivity | Day 1, Day 7 (8 hours post typhoid vaccine), Day 8 (32 hours post typhoid vaccine)
  Comparison of change in platelet reactivity from baseline after typhoid vaccination following nitrate versus placebo supplementation
Plasma nitrate concentration | Day 1, Day 7 (8 hours post typhoid vaccine), Day 8 (32 hours post typhoid vaccine)
  Comparison of change in plasma nitrate concentration following inorganic nitrate versus placebo supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Ahluwalia, BSc PhD, Principal Investigator — William Harvey Research Institute, Barts and The London, Queen Mary's School of Medicine and Dentistry
Locations (1):
- William Harvey Research Institute, Barts and The London School of Medicine, London, United Kingdom

REFERENCES:
- [Background] Hingorani AD, Cross J, Kharbanda RK, Mullen MJ, Bhagat K, Taylor M, Donald AE, Palacios M, Griffin GE, Deanfield JE, MacAllister RJ, Vallance P. Acute systemic inflammation impairs endothelium-dependent dilatation in humans. Circulation. 2000 Aug 29;102(9):994-9. doi: 10.1161/01.cir.102.9.994. PMID 10961963
- [Background] Kharbanda RK, Walton B, Allen M, Klein N, Hingorani AD, MacAllister RJ, Vallance P. Prevention of inflammation-induced endothelial dysfunction: a novel vasculo-protective action of aspirin. Circulation. 2002 Jun 4;105(22):2600-4. doi: 10.1161/01.cir.0000017863.52347.6c. PMID 12045164
- [Background] Donald AE, Charakida M, Cole TJ, Friberg P, Chowienczyk PJ, Millasseau SC, Deanfield JE, Halcox JP. Non-invasive assessment of endothelial function: which technique? J Am Coll Cardiol. 2006 Nov 7;48(9):1846-50. doi: 10.1016/j.jacc.2006.07.039. Epub 2006 Oct 17. PMID 17084260
- [Background] Clapp BR, Hingorani AD, Kharbanda RK, Mohamed-Ali V, Stephens JW, Vallance P, MacAllister RJ. Inflammation-induced endothelial dysfunction involves reduced nitric oxide bioavailability and increased oxidant stress. Cardiovasc Res. 2004 Oct 1;64(1):172-8. doi: 10.1016/j.cardiores.2004.06.020. PMID 15364625
- [Derived] Lau C, Primus CP, Shabbir A, Chhetri I, Ono M, Masucci M, Bin Noorany Aubdool MA, Amarin J, Hamers AJ, Khan Z, Kumar NA, Montalvo Moreira SA, Nuredini G, Osman M, Whitear C, Godec T, Kapil V, Massimo G, Khambata RS, Rathod KS, Ahluwalia A. Accelerating inflammatory resolution in humans to improve endothelial function and vascular health: Targeting the non-canonical pathway for NO. Redox Biol. 2025 May;82:103592. doi: 10.1016/j.redox.2025.103592. Epub 2025 Mar 28. PMID 40209616